CLINICAL TRIAL: NCT01476150
Title: Prevalence and Predictors of Osteoporosis in the Beijing's Urban Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Guochun Wang, Chief, Dept. of Rheumatology & Immunology, China-Japan Friendship Hospital, China-Japan Friendship Hospital
Other Study IDs: CJFSRI-OP
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — complete blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Dongcheng
- Haidian
- Xicheng
- Chaoyang
- Chongwen
- Tongzhou
- Fengtai
- Xuanwu

SUMMARY:
1. To establish a BMD reference database of Beijing's urban population, China.
2. To determine the prevalences and risk factors of osteoporosis and osteopenia in Beijing's urban population, China.
3. To describe the 25OHD level and estimate the prevalence of vitamin D insufficiency and deficiency of Beijing's urban population, China.
4. Estimation of the prevalence of osteoporotic fracture (vertebral) in over age of 60 of Beijing's urban population, China.

DETAILED DESCRIPTION:
With one of the biggest populations in the world, China was heavily suffered from osteoporosis. The prevalence of osteoporosis in China even is increasing fast in recent years, which are especially notable in urban population. This change maybe due to the conditions including rapid economic growth, increase in life expectancy, and changes in lifestyle. Studies in 1998 including 13 separately small samples (no more than 1000 people) from 9 provinces in China showed that the prevalence of osteoporosis and osteopenia were 5.3-6.2% and 5.8-11.2%, respectively. These estimates were higher by approximately 1% than those reported in 1995. In 2002, according to DEXA results in connection with population census in 2000, Xiaoguang Cheng et al. took a survey in 600 people who were separately studied in previously 10 research projects and find that patients with osteoporosis account for approximately 6.97% of the total China population.

Although these studies have documented a remarkable increase in the prevalence of osteoporosis in China, these estimations were all based on small samples. No risk factors related with osteoporosis and osteopenia, esp. hypovitaminosis D on osteoporosis and osteopenia, have been analyzed yet. So it is impossible to make any forecast of osteoporosis or give any instruction for intervention.

Thus this study designed to provide current and reliable data on the prevalence of osteoporosis and osteopenia and associated risk factors correlation coefficients in the Beijing's urban adult population.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 79 residents in urban Beijing, China.

Exclusion Criteria:

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will comprise 10,000 people aging from 20 to 79 residing in urban Beijing, China. All of them are members of Beijing Municipal Health Insurance (Beijing is a city that buy medical insurances for all of its residents).
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
A BMD reference database of Beijing's urban population, China. | 2 years

SECONDARY OUTCOMES:
The prevalences and risk factors of osteoporosis and osteopenia in Beijing's urban population, China. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shukun Yao, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China